CLINICAL TRIAL: NCT02650596
Title: Effects of Liraglutide on Left Ventricular Function in Chronic Heart Failure Patients With Type 2 Diabetes
Brief Title: Effects of GLP-1 on Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Yang (Other)
Responsible Party: Sponsor-Investigator, Shi Yang, director, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 301nlxnk
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Glucagon-Like Peptide 1; Liraglutide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 group (Experimental): drug: liraglutide (Novo Nordisk, Bagsværd, Denmark); the frequency: Subcutaneous liraglutide were taken daily; duration: 3 months. After admission, the patients were treated with 0.6 mg liraglutide once daily for 1 week, then 1.2 mg liraglutide for another 1 week, and then 1.8 mg liraglutide to the end.
  Interventions: Drug: GLP-1
- Control group (Placebo Comparator): drug: placebo (Novo Nordisk, Bagsværd, Denmark); the frequency: Placebo were taken daily; duration: 3 months. After admission, the patients were treated with 0.6 mg placebo once daily for 1 week, then 1.2 mg placebo for another 1 week, and then 1.8 mg placebo to the end.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLP-1 — Liraglutide were taken daily for 3 months
  Other Names: Liraglutide
  Arms: GLP-1 group
Drug: Placebo — Placebo were taken daily for 3 months
  Arms: Control group

SUMMARY:
The investigators planned to evaluate the effects of liraglutide on left ventricular function in chronic heart failure patients with type 2 diabetes.

DETAILED DESCRIPTION:
Heart failure (HF) is a major cause of morbidity and mortality world wide. Glucagon-like peptide-1 (GLP-1) is an incretin hormone that regulates plasma glucose, and has direct effects on the cardiovascular system. In our previous study, the GLP-1 analogue liraglutide could improve left ventricular function in patients with acute myocardial infarction. However, the effects of GLP-1 on chronic heart failure patients with type 2 diabetes remain unclear. The aim of this study was to evaluate the effects of liraglutide on left ventricular function in chronic heart failure patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure patients with type 2 diabetes (NYHA-class I, II or III) were eligible for the study

Exclusion Criteria:

* CHF (NYHA class IV)
* Type 1 diabetes
* Hospitalisation due to incompensated heart disease within 30 days prior to randomisation
* Myocardial infarction within the past 3 months before screening
* Coronary revascularisation within the past 3 months before screening
* Atrial fibrillation with ventricular frequency >100/min in rest
* ECG suggestive of malignant ventricular arrhythmia
* Prolonged QT-interval (>500 ms)
* Valvular heart disease
* Current myocardial or pericardial infection
* Obstructive hypertrophic cardiomyopathy
* Cancer unless in complete remission for ≥5 years
* Acute pancreatitis
* Compromised kidney function (eGFR <30 mL/min), dialysis or kidney transplantation
* History of thyroidea adenoma or carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fraction measured by 3D echocardiography | 3 months
  The primary efficacy endpoint was the effect of liraglutide on left ventricular ejection fractions (LVEF) measured by 3D echocardiography at 3 months.

SECONDARY OUTCOMES:
plasma NT-proBNP levels | 3 months
  a change in plasma NT-proBNP levels at 3 months after treatment
a change in 6-minute walk distance | 3 months
  The change in 6-minute walk distance at 3 months after treatment.
differences in the incidences of treatment-emergent adverse events | 3 months
  differences in the incidences of treatment-emergent adverse events at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Timmers L, Henriques JP, de Kleijn DP, Devries JH, Kemperman H, Steendijk P, Verlaan CW, Kerver M, Piek JJ, Doevendans PA, Pasterkamp G, Hoefer IE. Exenatide reduces infarct size and improves cardiac function in a porcine model of ischemia and reperfusion injury. J Am Coll Cardiol. 2009 Feb 10;53(6):501-10. doi: 10.1016/j.jacc.2008.10.033. PMID 19195607
- [Result] Chen WR, Shen XQ, Zhang Y, Chen YD, Hu SY, Qian G, Wang J, Yang JJ, Wang ZF, Tian F. Effects of liraglutide on left ventricular function in patients with non-ST-segment elevation myocardial infarction. Endocrine. 2016 Jun;52(3):516-26. doi: 10.1007/s12020-015-0798-0. Epub 2015 Nov 16. PMID 26573925
- [Result] Chen WR, Hu SY, Chen YD, Zhang Y, Qian G, Wang J, Yang JJ, Wang ZF, Tian F, Ning QX. Effects of liraglutide on left ventricular function in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention. Am Heart J. 2015 Nov;170(5):845-54. doi: 10.1016/j.ahj.2015.07.014. Epub 2015 Jul 26. PMID 26542491